CLINICAL TRIAL: NCT00226512
Title: Phase III Trial of a Non-myeloablative Preparative Regimen With Fludarabine and Busulfan With or Without Anti-lymphocyte Antibodies (Campath-1H or ATG) for Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome Undergoing Allogeneic Stem Cell Transplantation From an HLA Compatible Donor
Brief Title: To Determine the Role of Adding Campath-1H or ATG Given In-vivo in Addition to Fludarabine and Low Dose Busulfex on Outcome in Patients Treated With Reduced Intensity Conditioning
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230704-HMO-CTIL
Record Dates: First submitted 2005-09-09; First posted 2005-09-27 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Alemtuzumab

INTERVENTIONS:
Drug: Campath-1H /ATG

SUMMARY:
Multi-institutional randomized phase III trial of a non-myeloablative preparative regimen with fludarabine and busulfex with or without anti-lymphocyte antibodies (monoclonal humanized Campath-1H administered s.c. or polyclonal rabbit anti-T lymphocyte antibodies (ATG), combined with low dose and short course cyclosporine A (CSA) and methotrexate (MTX) as the sole agent for prevention of graft-vs-host disease (GVHD) for patients with acute myelogenous leukemia or myelodysplastic syndrome undergoing allogeneic stem cell transplantation from an HLA compatible donor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML or MDS, with no lower or upper age limit:
* a) Induction failure
* b) First or subsequent remission
* c) Untreated first relapse
* Patients must have an HLA compatible donor willing and capable of donating peripheral blood stem cells (first choice) or bone marrow progenitor cells using conventional techniques and blood lymphocytes if indicated (HLA compatible defined as 5/6 or 6/6 matched related or 10/10 molecular matched unrelated donor (A,B,C,DR,DRB1).

Exclusion Criteria:

* Donor contraindication (HIV seropositive confirmed by Western Blot, Hepatitis B antigenemia).
* Evidence of bone marrow disease.
* Unable to donate bone marrow or peripheral blood due to concurrent medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2004-07

PRIMARY OUTCOMES:
To determine the efficacy of s.c. Campath-1H or ATG in decreasing the incidence and severity of acute and chronic GVHD in patients with AML and MDS treated with non-myeloablative stem cell transplantation.

SECONDARY OUTCOMES:
Investigate the role of different conditioning regimens on:
Infection, engraftment relapse rate and disease free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel